CLINICAL TRIAL: NCT06980441
Title: Feasibility and Acceptability of Culturally Adapted, Evidence-Informed Psychological Support on Mental Health Symptoms and Violence for Conflict-Affected Populations in Afghanistan: A Study Protocol
Brief Title: Culturally Adapted Psychological Support for Conflict-Affected Afghans: Study Protocol on Mental Health & Violence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peace of Mind Association (PoMA) (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Lyla Schwartz, Directors of Programs and Psychology, Peace of Mind Association (PoMA)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1378139
Record Dates: First submitted 2025-05-01; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Depression and Suicide Ideation; Anxiety; PTSD
Keywords: Youth mental health; Afghanistan; Implementation science; Culturally adapted psychological support; Evidence informed interventions; Mental health symptoms; Psychological experiences
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: PM+ EP (Experimental): Participants in this group will receive a culturally adapted version of the World Health Organization's Problem Management Plus (PM+) program, with an added Emotional Processing (EP) module. The intervention will be delivered through six individual sessions over one month by trained Afghan facilitators of the same gender as the participant. Sessions will focus on managing distress, solving problems, building social support, and processing difficult emotions.
  Interventions: Behavioral: Problem Management Plus with Emotional Processing module
- No Intervention Arm (No Intervention): Participants in this group will not receive the intervention during the study period but will complete the same assessments as the intervention group. After the study concludes, they will be offered the opportunity to receive the PM+ EP sessions.

INTERVENTIONS:
Behavioral: Problem Management Plus with Emotional Processing module — PM+ EP comprises of Problem Management Plus, an evidence-based low intensity psychological intervention developed by the World Health Organization (WHO), with an additional Emotional Processing module specifically to address psychological distress related to trauma exposure. The core of the intervention is designed for adults impaired by distress in communities exposed to conflict and adversity; it consists of CBT techniques that have been adapted for communities that do not have good availability of specialist care. The additional module was developed by researchers treating refugee youth (Alozkan Sever et al, 2021). For this study, PM+ EP will be a six-session individual and guided support program. The original sections of PM+ are available in many languages including Farsi, and the additional EP module will be translated by PoMA's Afghan translator. The sessions cover the topics of managing stress, strengthening social support, staying well and persevering.
  Arms: Intervention Arm: PM+ EP

SUMMARY:
This pilot study examines the feasibility and acceptability of a culturally adapted psychological intervention-Problem Management Plus with Emotional Processing (PM+ EP)-for young Afghans aged 16-30 experiencing high psychological distress. Through a pilot randomized control trial and qualitative interviews, the study explores whether PM+ EP can reduce symptoms of anxiety, depression, PTSD, and aggression, and improve daily functioning. Findings will inform the potential for a larger trial and address critical mental health and violence prevention needs in conflict-affected Afghan communities.

DETAILED DESCRIPTION:
Background: A large portion of Afghanistan's population, particularly children, has endured prolonged conflict, poverty, and displacement, leading to significant psychological distress. As children grow into adolescence and adulthood, this distress often manifests in mental health symptoms and an increased likelihood of violent behaviours. With limited mental health professionals and strong stigma around mental health in Afghanistan, culturally adapted, evidence-based interventions are needed.

Objective: The study aims to explore the feasibility and acceptability of culturally adapted mental health intervention Problem Management Plus with an additional Emotional Processing module (PM+ EP), in reducing psychological distress in young Afghans. The primary objective is to assess the feasibility of delivering this intervention in Afghanistan and its acceptability by the target communities, and the secondary objective is to assess symptom reduction and behavioural change.

Methods: This is a pilot Randomized Control Trial (RCT) with participants aged 16 to 30 in Afghanistan. Eligible participants, young Afghans with high levels of distress and impaired functioning - measured by the Kessler Psychological Distress Scale (K10) -, will be randomized to PM+ EP (n=30) or the waiting group (n=30). The participants will be evaluated through self-report questionnaires at three time points; baseline (T1), four weeks later immediately post-intervention (T2), and 3 months post-intervention (T3), and through a qualitative interview (Process Evaluation) at the end of the study. Outcomes will include measures of anxiety and depression (HSCL-25), aggressive behaviours (AGQ), PTSD symptoms (PCL-5), and daily functioning (WHODAS 2.0).

Analysis: This study will assess the feasibility and acceptability of culturally adapted PM+ EP in Afghanistan and explore the relationship between mental health symptoms and violence among young Afghans. It will be the first to evaluate the feasibility of PM+ EP with this population and could pave the way for a large define RCT examining the effectiveness this approach, should the results show promise.

ELIGIBILITY:
Inclusion Criteria:

* Psychological Distress, measured at >15 on the Kessler Psychological Distress Scale (K10)
* Afghan nationality
* Age between 16 and 30
* Ability to read and write in Dari

Exclusion Criteria:

* Imminent suicide risk
* Experiencing psychosis
* Neurological or cognitive disabilities

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in psychological distress symptoms among participants, as measured by scientific scale HSCL-25. | Pre-intervention until 3 months post-intervention
  In this pilot RCT, the primary outcome is to explore the feasibility and acceptability of delivering the PM+ EP intervention in Afghanistan. The study serves to demonstrate whether such interventions could be safety scaled and produce positive outcomes for the target population. All participants will complete four surveys for assessment at study points T0, T1, T2 and T3. The Hopkins Symptom Checklist 25 (HSCL-25) is one outcome measure designed to measure for anxiety and depression. Hopkins Symptom Checklist-25 (HSCL-25) is a 25 item self-report questionnaire assessing symptoms of psychological distress; 10 items for anxiety symptoms and 15 items for depression symptoms (2 of which identify somatic symptoms) (Mollica et al, 1987). The items are rated on a 4-point Likert scale, ranging from 1 (never) to 4 (always) with the anxiety scale ranging from 10-40 and the depression scale from 15-60. The total scale (range 25-100) represents psychological distress.
Reduction in psychological distress symptoms among participants, as measured by scientific scale DSM-5 (PCL-5). | Pre-intervention until 3 months post-intervention
  The primary outcome of this pilot RCT is to assess the feasibility and acceptability of delivering the PM+ EP intervention in Afghanistan and its potential for safe scale-up and positive impact. All participants will complete four assessments at T0, T1, T2, and T3. PTSD symptoms will be measured using the PTSD Checklist for DSM-5 (PCL-5), a 20-item self-report tool that assesses symptoms over the past month. Each item is scored from 0 (Not at all) to 4 (Extremely), covering four symptom clusters: Re-experiencing, Avoidance, Negative Cognition/Mood, and Hyperarousal. A provisional PTSD diagnosis can be made if participants endorse the minimum number of symptoms in each cluster at a rating of 2 or higher. A total score between 31-33 suggests probable PTSD. This outcome will help determine whether PM+ EP is a feasible and acceptable approach to reducing trauma symptoms among conflict-affected youth in Afghanistan.
Reduction in psychological distress symptoms among participants, as measured by scientific scale WHODAS 2.0. | Pre-intervention until 3 months post-intervention
  The primary outcome of this pilot RCT is to assess the feasibility and acceptability of delivering the PM+ EP intervention in Afghanistan, evaluating its potential for safe scale-up and positive outcomes. All participants will complete four assessments at T0, T1, T2, and T3. Functional ability will be measured using the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0), a validated tool developed by WHO to assess health and disability across six domains: cognition, mobility, self-care, getting along, life activities, and participation. Participants report difficulties experienced in the past 30 days on a five-point Likert scale (1 = none to 5 = extreme), with total scores ranging from 12 to 60. Higher scores indicate greater functional impairment. This outcome will inform whether PM+ EP is feasible, acceptable, and functionally beneficial for young Afghans experiencing psychological distress.

SECONDARY OUTCOMES:
Participant-Reported Changes in Attitudes Toward Violence and Perceived Impact of PM+ EP on Mental Health and Behavior. | 3 months post-intervention
  This outcome explores the relationship between mental health symptoms and violent behavior through qualitative interviews with a purposive sample of participants and facilitators conducted after the intervention (T3). Interviews will investigate perceived changes in psychological distress, aggressive behavior, and attitudes toward violence, as well as the cultural relevance and acceptability of the PM+ EP intervention. Data will be analyzed thematically using ATLAS.ti. Results will be used to illustrate context-specific linkages between mental health and violence and to inform future adaptation and scale-up of culturally tailored psychological interventions in conflict-affected settings.
Analysis of relationship between mental health and violence, as measured by scientific scale AGQ. | Pre-intervention until 3 months post-intervention
  The study's secondary outcome is to examine the relationship between mental health and violence, and assess the potential impact of culturally adapted mental health programming on symptom and behavioral change, particularly in reducing violence. Aggression will be measured using the Aggression Questionnaire (AGQ), a 29-item self-report tool assessing physical aggression, verbal aggression, anger, and hostility. Participants rate each item on a 7-point Likert scale (1 = extremely uncharacteristic of me; 7 = extremely characteristic of me), with total scores ranging from 29 to 203. Higher scores indicate greater levels of aggression. The AGQ captures both aggressive acts and temperamental traits, allowing for analysis of change in aggressive behaviors and attitudes over time. This outcome will contribute to understanding context-specific linkages between mental health symptoms and violence in conflict-affected populations.

CONTACTS AND LOCATIONS:
Overall Officials: Lyla L Schwartz, Masters, Principal Investigator — Peace of Mind Association (PoMA)
Locations (1):
- Peace of Mind Association (PoMA), Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data will be available upon request after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted immediately after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and the signing of a Data Sharing Agreement (DSA).

DOCUMENTS (1):
  • Study Protocol (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT06980441/Prot_000.pdf